CLINICAL TRIAL: NCT03548883
Title: Examining Neuroinflammation in AlzHeimer's Disease Via TrAnscriptomic ProfiliNg and MiCroglia ModEling Using Human Peripheral Blood Mononuclear Cells (ENHANCE)
Brief Title: Examining Neuroinflammation in AlzHeimer's
Acronym: ENHANCE
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 864676
Record Dates: First submitted 2017-02-13; First posted 2018-06-07 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease, Early-Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
  Materials of human origin will be collected in the manner described in the specific study visits. Testing that is not conducted at FH will be conducted at SBP, University of Miami or other collaborating laboratories. A Material Transfer Agreement will be obtained, which will govern the transfer of tissue and the chain of custody of the tissue outside of FH for this endpoint testing. If any requests are received from an outside entity for archived tissue, a Material Transfer Agreement will be obtained, which will govern the transfer of tissue and the use of the tissue outside of FH.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Alzheimer subject Group: In phase I, up 50 AD patients will be recruited and screened until we obtain 6 AD subjects. All potential subjects recruit will be pre-screened for initial inclusion/exclusion criteria via examination of standard of care (SOC) medical history, labs, imaging, and cognitive assessment. Recruited subjects will be scheduled for Study Visit #1 (@TRI) and will be further screened with protocol cognitive assessments, depression screening, assessment of daily activities, and labs. During Study Visit #2, these subjects will undergo structural imaging with high resolution magnetic resonance imaging (@ TRI) without contrast (MRI), to rule out other causes of cognitive decline.
- Control Group: In phase II, up to 50 age, sex, race ethnicity, group matched healthy controls will be recruited and screened until we have 6 healthy control subjects. All potential subjects recruit will be pre-screened for initial inclusion/exclusion criteria via examination of medical history (including a review of past images, current medication and labs if available). Recruited subjects will be scheduled for Study Visit #1 and will be further screened with protocol cognitive assessments, depression screening, assessment of daily activities, and labs. During Study Visit #2, these subjects will undergo structural imaging with high resolution magnetic resonance imaging (@ TRI) without contrast (MRI), to confirm that there are no undiagnosed conditions.
- Type 2 diabetes group: In phase III, up to 50 age, sex, race ethnicity, group matched T2D patients will be recruited and screened until we have 6 T2D subjects. All potential subjects recruit will be pre-screened for initial inclusion/exclusion criteria via examination of medical history (including a review of past images, current medication and labs if available). Recruited subjects will be scheduled for Study Visit #1 and will be further screened with protocol cognitive assessments, depression screening, assessment of daily activities, and labs. During Study Visit #2, these subjects will undergo structural imaging with high resolution magnetic resonance imaging (@ TRI) without contrast (MRI), to confirm that there are no undiagnosed conditions.

SUMMARY:
Alzheimer disease (AD) is a neurodegenerative disorder with a poorly understood pathology. It is an irreversible progressive brain disease that slowly deteriorates memory, thinking and behavior. It affects the elderly population and is also hereditary. The incidence doubles with every decade after sixty with no signs of leveling off. More than 35 million people Worldwide, including 5.5 million living in the United States, suffer from AD. As the United States population ages, it is expected that the number of people with AD will increase, reaching 13.2 to 16.0 million by the year 2050. The cost of care for patients with AD in the United States is expected to rise as well, from $172 billion a year in 2010 to a trillion dollars a year by 2050.

Although the exact etiopathology is not known there are several lines of evidence that suggest that metabolic and inflammatory features are important. It also has been known for many years that the Blood Brain Barrier (BBB) of Alzheimer's patients allow more harmful particles to cross into the brain than the BBBs of those without the disease do. It's known that this barrier, which is regulating transfer of molecules between the brain and blood, and vice versa blood and brain, can become leaky and dysfunctional (in particular capillaries dysfunction) and lead to subsequent problems likely contributing to onset and progression of dementia. This protocol will explore several of the most promising putative factors that cause AD.

ELIGIBILITY:
INCLUSION criteria AD Subject Group:

* Age ≥ 60
* Subject must have a diagnosis of AD by a licensed neurologist, psychiatrist, or geriatrician
* Subject must have mild to moderate AD as determined by cognitive or behavioral symptoms that interfere with functioning in usual daily activities found in the medical history and/or demonstrated by the following assessments results:
* Mini Mental Status Examination (MMSE) score of 12≤x≤24
* Alzheimer's Disease Assessment Scale ADAS-cog score of 18≤x≤37
* Clinical Dementia Rating (CDR) Score of 1 or 2
* Blessed Dementia Scale (Activities of Daily Living) Score of 1≤x≤11
* Under Changes in Performance of Everyday Activity
* Subject/LAR cannot report severe loss (score of 1) in the following categories because it indicates severe dementia:

Inability to find way about indoors (home or familiar location) Inability to interpret surroundings, for example, to recognize whether in hospital or home, etc.

Under Changes in Habit

* Subject/LAR cannot report severe loss (score of 3) in any of the following categories because it indicates severe dementia Eating Dressing Sphincter control No history of neurological or non-neurological conditions that cause cognitive impairments found in physician notes and/or CT or MRI results (from medical history or protocol MRI)such as Dementia with Lewy bodies Frontotemporal dementia History of strokes in which the patient did not return to previous level of activity and cognition Seizure History in which the patient had residual cognitive deficits Presence of multiple or extensive infarcts or severe white matter hyper-intensity burden Subjects with history of head trauma will be reviewed by PI and Sub-Is and will be included or not at the their discretion.
* No history psychiatric diagnosis that predates AD diagnosis by 3 years or more
* No active delirium Assessed by the Confusion Assessment Method (CAM). Subject will be considered positive for delirium if patient has presence of features 1 and 2 and either 3 or 4
* Individuals willing and able to sign the informed consent either by themselves or with the assistance of an interpreter or legally authorized representative
* Individuals capable of having an MRI with contrast
* A score in the normal or mild depression range (0 to 19 on the Geriatric Depression Scale

INCLUSION criteria Healthy Control and Type 2 Diabetes (T2D) Subject Groups:

* Volunteers who are ≥ 60 and age (±5years), sex, race, and ethnicity matched to participating AD subjects
* No self-reported or document medical history of current or prior psychiatric, neurological, or non-neurological conditions that cause cognitive impairments, such as Lewy bodies, or other conditions the PI thinks would impact the study results, found in physician notes CT or MRI results (from medical history or protocol MRI)
* Subjects with history of head trauma will be reviewed by PI and Sub-Is and will be included or not at the their discretion. Subjects with history of strokes in which the patient did not return to previous level of activity and cognition will be excluded. If a subject with a previous stroke returned to the baseline, the subject can be included in the study.
* History of seizure in which the patient had residual cognitive deficits. If subject seizure history did not result in cognitive impairments the subject can be included
* Mini Mental Status Examination (MMSE) score of x≥25
* Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog) score of 18≥x
* Blessed Dementia Scale (Activities of Daily Living) Score of 0
* Clinical Dementia Rating (CDR) Score of 0
* No history of psychiatric diagnosis
* No active delirium
* Subjects will be considered positive for delirium if patient has presence of features 1 and 2 and either 3 or 4
* A score in the normal range (0 to 9) on the Geriatric Depression Scale Individuals willing and able to sign the informed consent by themselves Individuals capable of having an MRI with contrast

INCLUSION criteria T2D Subject Group:

* Glycosylated hemoglobin (Hba1c) ≥ 7.5%
* For subjects who are treated with glucose lowering medications, should be controlled (defined as HbA1c ≤ 9.5%) on a stable dose of medications for at least 3 months prior to screening.

EXCLUSION criteria for AD Subject , Healthy Control Subject and T2D Subject Groups:

* Age ≤ 60
* Unable/Does not wish to provide blood sample
* Unable to have MRI with and without contrast to exclude other diagnoses
* Patient who is allergic
* Patient who requires sedation for any reason/unable to tolerate MRI imaging ( ex.(ex. claustrophobia, or anxiety)
* Past or current medical history of psychiatric or neurological conditions that cause cognitive impairments, such as Lewy bodies, stroke, seizure, any other medications PI thinks would impact the study results.
* Subjects with history of head trauma will be reviewed by PI and Sub-Is and will be included or not at the their discretion.
* Subjects with history of strokes in which the patient did not return to previous level of activity and cognition will be excluded. If a subject with a previous stroke returned to their baseline the subject can be included in the study.
* History of seizure in which the patient had residual cognitive deficits. If subject seizure history did not result in cognitive impairments, the subject can be included
* Research team has the right to exclude any subjects based on any findings that might impact the subjects ability to participate in the study
* Active delirium (Subjects will be considered positive for delirium if patient has presence of features 1 and 2 and either 3 or 4)
* Abnormal results indicated the possibility of secondary cause of dementia such as Vitamin B12 deficiency, hypothyroidism, hypoparathyroidism, anemia, hypoxia, or hypercapnia, hepatic and renal encephalopathies, and dehydration would make the subject a screen failure. Specifically:
* Liver disease (AST or ALT >2.5 times the upper limit of normal)
* Anemia (hemoglobin <12 g/dl in men, <11 g/dl in women)
* Thyroid dysfunction (TSH below the lower limit of normal; TSH above the upper limit of normal if symptomatic; TSH >10 mIU/L if symptomatic or asymptomatic); if TSH above the upper the limit of normal and ≤10 mIU/L, subject will be informed about the finding to make a decision on whether or not to participate in the study, which will be recorded in the subject's medical record.
* History of diabetes type I
* History of diabetes type II with HbA1c >7.5%
* Erectile dysfunction drugs (If subject can stop taking erectile dysfunction drug for 2 weeks prior to study participation and remain off the drug through Study Visit #2 participation, the subject can be enrolled)
* Acute or chronic severe renal insufficiency (glomerular filtration rate < 30 mL/min/1.73m2); or renal dysfunction due to the hepato-renal syndrome or in the perioperative liver transplantation period. In the hepato-renal syndrome or in the perioperative liver transplantation period, the risk applies to any severity of renal dysfunction.
* Uncontrolled hypertension (BP > 140 systolic or 90 diastolic). Will rescreen if controlled and patients can return for a second screening be reviewed by PI/Sub-I (assessing incidences of White Coat Syndrome). Inclusion in the study will be at the discretion of the PI.
* Patients taking anti-hypertensive medications will be excluded if the eGFR is <40ml min/1.73 m2 [28]. (eGFR will be calculated as per MDRD equation: eGFR (mL / min/1.73 m2) = 175 × (serum creatinine in mg/dl)-1.154 × (age in years)-0.203 ×(0.742 if female) × (1.212 if African American) or Updated Schwartz equation: eGFR (mL / min/1.73 m2) = (0.413 × height in cm)/serum creatinine in mg/dl. Patients with eGFR of > 40ml min/1.73 m2 will be included in the study. For GFR < 60 and >40 oral hydration is recommended, to consist of at least 500 ml (i.e. 2 cups) before contrast administration. We will follow the recommendation.
* Use of oral contraceptives or hormone replacement therapy.
* History of drug or alcohol abuse (> 3 drinks per day) in the last 5 years, or psychiatric disease prohibiting adherence to study protocol.
* History of cancer that is still ongoing. If cancer has been resolved, patient can be enrolled
* History of organ transplant.
* History of HIV, active Hepatitis B or C, or Tuberculosis.
* History of myocardial infarction within the past 6 months.
* Presence of clinically significant abnormalities on EKG.
* Current smokers (smoking within the past 3 months)
* Medication history will be taken and medications included or not at the PI's discretion.

EXCLUSION criteria only for AD Subject Group:

- If in the medical history, the subject's geriatrician, psychiatrist, or neurologist indicates that the subject has severe or advanced AD (not mild or moderate AD) and/or if the subject scores the following on Visit #1 assessments: Subject scores x≤18 and x≥37on the ADAS-cog Subject scores x≤12 and x≥24 and on the MMSE Subject scores 0 or x≥11 and on the Blessed Dementia Scale Subject scores x=0,0.5,or 3 and on the Clinical Dementia Scale

* Subject's MRI indicates any comorbid neurological or non-neurological conditions that could have a substantial effect on cognition. In the event that AD subject MRI indicates any comorbid neurological or non-neurological conditions, the subject will be considered a screen failure
* Use of narcotic medication that could have substantial effect on cognition
* History of psychiatric diagnosis that predates AD diagnosis by 3 years or more
* Subject scores above mild depression x > 19 on the GDS scale

EXCLUSION criteria only for control Subject and T2D Subject Groups:

* Subject scores ≥18 on ADAS-Cog (cognitive assessment).
* Subject's MRI indicates neurological or non-neurological conditions that could have a substantial effect on cognition. In the event that AD subject MRI indicates any neurological or non-neurological conditions that could have a substantial effect on cognition, the subject will be considered a screen failure and referred for medical evaluation.
* Subjects unable to sign consent themselves
* History of psychiatric diagnosis
* Use of medication that could have substantial effect on cognition: Psychoactive, Narcotic, Long-acting benzodiazepines, Anticonvulsants, Histamine H2 Receptor antagonist (Ex. Stimulants, Depressants, , Hallucinogens, Cannabis, Xanax, CodeinCodeine, Zyrtec, Zantac, Pepcid, Neurontin, Depakote, Depakene any other medications PI thinks would impact the study results)
* Subject scores above normal x > 9 on the GDS scale

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The team will have 12 AD patients for phase III. The team will have 12 healthy age and sex match controls for phase III.
  Due to the target study population, patients with AD, it is expected that the subjects will have cognitive impairments. The objectives of this study cannot be met with research only involving subjects who can personally give consent. Patients with AD who have cognitive impairments would have to be included in this study in order for us to accurately study the disease. For this study, a score of 24 or below on the Mini Mental Status Examination (MMSE), will indicate cognitive impairment. In these cases, we will get written consent from the legally authorized representative (LAR).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Compare the Blood Brain Barrier leaking between AD, T2D and healthy control subjects. | Two years
  A MRI of the brain with contrast will be used to assess the permeability of the Blood Brain Barrier.
Age | Two years
  Measured in years
Gender | Two years
  (Male or Female)
Body composition | Two years
  Measured by Dexascan
Weight | Two years
  Measured in kilograms
Height | Two years
  Measured in meters
BMI | Two years
  will be determined by dividing weight by height (square)
Race | Two years
  White/Black or African American/Asian/Other/Unknown or not reported
Cognitive data | Two years
  Evaluated by ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) questionnaire. Total scoring range of 0 - 70.
  The ADAS score is based on the number of errors made in each item. A score of 70 represents the most severe impairment and 0 represents the least impairment.
Lipid profile | Two years
  Measured of the HDL, LDL and VLDL content in the blood (measured in mg/dL)
Insulin | Two years
  Measured of insulin level in the blood
Adiponectin | Two years
  Measured of adiponectin level in the blood
Free Fatty Acid | Two years
  Measured of free fatty acid level in the blood
Transcriptomic profiles of the cells isolated from the blood | Two years
  after isolation of the peripheral blood mononuclear cell (PBMC) from the blood, measure of gene expression by RT-qPCR (real time quantitative polymerase chain reaction)
Activity monitoring - energy cost of free-living activity | Two years
  measured by wearing an arm band - measured in minutes
Epigenetic | Two years
  after isolation of the PBMC from the blood measure of DNA methylation
Metabolic of the cells isolated from the blood | Two years
  after isolation of the PBMC from the blood measure of metabolites by MS
Proteomic of the cells isolated from the blood | Two years
  after isolation of the PBMC from the blood, measure of proteins by western blot
Activity monitoring - lying down time | Two years
  measured by wearing an arm band - measured in minutes
Activity monitoring - sleeping time | Two years
  measured by wearing an arm band - measured in minutes
Cognitive data | Two years
  Evaluated by Clinical Dementia Rating (CDR) questionnaire
Cognitive data | Two years
  Evaluated by the Mini Mental Status Exam (MMSE)
Cognitive data | Two years
  Evaluated by the Blessed Dementia Scale (BDS) questionnaire
Cognitive data | Two years
  Evaluated by the Confusion Assessment Method (CAM)
Cognitive data | Two years
  Evaluated by the Geriatric Depression Scale (GDS)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Smith, MD, Principal Investigator — Florida Hospital Translation Research Institute

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ballard C, Gauthier S, Corbett A, Brayne C, Aarsland D, Jones E. Alzheimer's disease. Lancet. 2011 Mar 19;377(9770):1019-31. doi: 10.1016/S0140-6736(10)61349-9. Epub 2011 Mar 1. PMID 21371747
- [Result] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Result] Wang J, Yu JT, Tan MS, Jiang T, Tan L. Epigenetic mechanisms in Alzheimer's disease: implications for pathogenesis and therapy. Ageing Res Rev. 2013 Sep;12(4):1024-41. doi: 10.1016/j.arr.2013.05.003. Epub 2013 May 17. PMID 23688931
- [Result] Maiese K. "Connecting the dots" from blood brain barrier dysfunction to neuroinflammation and Alzheimer's disease. Curr Neurovasc Res. 2014;11(3):187-9. doi: 10.2174/1567202611666140609144347. No abstract available. PMID 24909964